CLINICAL TRIAL: NCT07228208
Title: Role of Endothelial Dysfunction on Exercise Pressor Reflex in Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, William Hughes, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO00053449
Record Dates: First submitted 2025-11-05; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes (T2DM); Endothelial Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either active or placebo supplement, acting as their own control
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant Supplementation (Experimental): MitoQ, a mitochondrial target antioxidant, given once at a dose of 160 mg
  Interventions: Dietary Supplement: MitoQ (mitoquinol mesylate)
- Placebo (Placebo Comparator): A placebo similar visually will be used to compare to MitoQ
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MitoQ (mitoquinol mesylate) — During each testing session, the investigators will be measuring how one treatment of an over-the-counter antioxidant supplement affects blood flow and muscle function. One day participants will orally ingest an over-the-counter antioxidant supplement called MitoQ.
  Arms: Antioxidant Supplementation
Dietary Supplement: Placebo — During each testing session, the investigators will be measuring how one treatment of an over-the-counter antioxidant supplement affects blood flow and muscle function. One day participants will orally ingest an over-the-counter antioxidant supplement called MitoQ, while the other they will ingest a placebo
  Arms: Placebo

SUMMARY:
Exaggerated blood pressure responses to exercise in individuals with Type 2 Diabetes significantly increase the risk of heart attack, stroke, and cardiovascular death, while also limiting exercise capacity and therapeutic benefits of physical activity. This research will determine whether impaired blood vessel function and excessive cellular damage from oxygen-containing molecules cause these dangerous blood pressure responses during exercise. The findings will establish whether targeting cellular antioxidant systems represents a new therapeutic approach to improve exercise tolerance and reduce cardiovascular risk in t Americans living with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes: 18 - 80 years old, able to give informed consent, > 6 months post-diagnosis, > 6 months stable medications for management
* Healthy controls: 18 - 80 years old, able to give informed consent

Exclusion Criteria:

* Type 2 Diabetes: Type 1 diabetes, symptomatic coronary artery disease, cardiovascular event in last year (MI, stroke), uncontrolled or unmanaged hypertension (>160/90 mmHg), heart failure, renal impairments, current or recent (<6 months) tobacco use, hormone replacement therapy, documented neuromuscular disorders, pregnancy
* Healthy Controls: Same as listed in Type 2 Diabetes with Type 2 Diabetes as an exclusion factor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure | Prior to and 45 minutes following supplement
  Change in mean arterial pressure is measured in response to handgrip exercise and post-exercise circulatory occlusion
Heart Rate | Prior to and 45 minutes following supplement
  Change in heart rate is measured in response to handgrip exercise and post-exercise circulatory occlusion

SECONDARY OUTCOMES:
Brachial Artery FMD | Prior to and 45 minutes following supplementation
  Brachial artery FMD a measure of endothelial function will be measured on the non-dominant arm
Plasma MitoQ Concentration | Prior to and 45 minutes following supplementation
  Circulating concentrations of MitoQ is assessed in blood via venipuncture
Muscle Tissue Oxygenation | Prior to and 45 minutes following supplementation
  We will also place a near-infrared spectroscopy (NIRS) pad on the thenar eminence of the non-paretic hand to non-invasively measure tissue oxygenation via infrared light following the pneumatic forearm cuff inflation/deflation.

CONTACTS AND LOCATIONS:
Overall Officials: William E Hughes, Ph.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No